CLINICAL TRIAL: NCT06200792
Title: The Impact of Stress in Residents' Performance
Brief Title: Stress and Anxiety Affect Residents' Performance
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Principal investigator, University of Padova
Other Study IDs: Stress study
Record Dates: First submitted 2023-12-07; First posted 2024-01-11 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Stress; Stress Disorder; Work Related Stress
MeSH Terms: conditions — Stress Disorders, Traumatic; Occupational Stress | interventions — Surveys and Questionnaires; Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: eSense device — eSense device for monitoring electrodermal activity. Visual analogic scale (VAS) for pain and discomfort; TOL-R tests for investigating working performances.
  Other Names: Questionnaires and scales for evaluating esecutive function.

SUMMARY:
Being an anesthesiologist implies huge dedication and both physical and psychological efforts. None has ever studied the impact of a working day on anxiety, perceived stress levels, physiological data, and executive functions.

DETAILED DESCRIPTION:
During a working day, trainees will have their physiological and psychological data recorded before starting their clinical activity and after them. Electrodermal activity with the eSense device, Executive functions through the TOL-R and all the questionnaires and scales will be sampled at the beginning of the day and at the end of the day the same procedure will be applied again (exclusion for PSS-10 scale, STAY-Y trait anxiety and GAD-7) eSense and TOL-R, are useful tools to understand sympathetic activity and executive functions. The galvanometer it is the gold standard to measure EDA; i.e. electrodermal activity, which is a pure sympathetic index, while Tower of London it is the gold standard to assess planning, monitoring and programming skills, both data are supposed to be heavily involved in an anesthesiologist trainee during the all day.

The aims of the study are to evaluate executive functions at the start and at the end of a working day and to understand theirs relationship with anxiety, perceived stress levels and physiological changes in sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* Being an anesthesiologist residents
* Written informed consent obtained

Exclusion Criteria:

* Psychiatric disorders
* Neurological disorders
* Suffering from high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anesthesiologists residents
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Differences in executive functions overtime | baseline and immediately after intervention
  Evaluating executive functions at the start and at the end of a working day using the Tower of London test (TOL-R) (scoring 0 (worst score)-30 (better score))

SECONDARY OUTCOMES:
Differences in dermal activity during working day | baseline and immediately after intervention
  Evaluating potential differences in electrodermal activity overtime using microsiemens, counting number of stress response
Assess the general level of anxiety | baseline and immediately after intervention
  Measuring levels of anxiety using the generalized anxiety disorder-7 item (GAD-7) (minimum 0, maximum score 21)
General level of anxiety | baseline and immediately after intervention
  Measuring the general levels of anxiety with the Stait-trait anxiety inventory (STAI-Y1-2) (1 point=not at all/almost never anxiety; 2=somewhat/sometimes; 3=moderately so/often) and 4= very much so/almost always)
Evaluating the general levels of perceived stress levels | baseline and immediately after intervention
  Evaluation of the general levels of perceived stress levels using the perceived stress score (PSS)-10 scale (0 (minimum level of anxiety)-10 (maximum level of anxiety))

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontoiatrica, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
Nope